CLINICAL TRIAL: NCT00841308
Title: Antihypertensive Drug Treatment Decisions Based on Home Blood Pressure Monitoring
Brief Title: Home Blood Pressure in Hypertension Management
Acronym: HBP10
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, George S. Stergiou, Associate Professor of Medicine and Hypertension, University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HBP10
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator)
  Interventions: Other: Decision to start and titrate drug treatment based only on home blood pressure monitoring
- Home blood pressure monitoring (Active Comparator)
  Interventions: Other: Decision to start and titrate drug treatment based only on home blood pressure monitoring

INTERVENTIONS:
Other: Decision to start and titrate drug treatment based only on home blood pressure monitoring — Drug Treatment according to current Hypertension Guidelines. Decision to start and titrate drug treatment based on clinic and ambulatory blood pressure ("Usual care" arm) versus based on home blood pressure monitoring only ("Home blood pressure monitoring" arm).

SUMMARY:
This is a prospective randomized study with two arms: the Conventional and Ambulatory blood pressure monitoring arm and the Home blood pressure monitoring arm. The study will include both previously treated and untreated individuals.

Before randomization and in the end of the study, measurements will be performed using all three blood pressure monitoring methods (Conventional, Ambulatory and Home) as well as assessment of target organ damage (microalbuminuria, electrocardiogram, echocardiogram, carotid-femoral pulse wave velocity and central blood pressure).

The participants will be randomized into one of the two arms. Diagnosis and titration will be decided according to either Conventional and Ambulatory blood pressure measurements or according to Home blood pressure measurements. Subjects will be followed up for one year.

ELIGIBILITY:
Inclusion Criteria:

* Untreated hypertensive adults
* Treated hypertensive adults with uncontrolled blood pressure

Exclusion Criteria:

* Stage III Hypertension
* Secondary Hypertension
* Cardiovascular or Renal disease
* Uncontrolled Diabetes

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-02; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Intermediate target organ damage (Left Ventricular Hypertrophy, Microalbuminuria, carotid-femoral Pulse Wave Velocity, Central blood pressure) | Baseline and 12 months

SECONDARY OUTCOMES:
Blood Pressure Control, Cost-Effectiveness | Baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: George S Stergiou, MD, Study Chair — Hypertension Center, Third Depertment of Medicine, University of Athens, Greece
Locations (1):
- Hypertension Center, Third Department of Medicine, University of Athens, Greece, Athens, Greece

REFERENCES:
- [Derived] Nasothimiou EG, Karpettas N, Dafni MG, Stergiou GS. Patients' preference for ambulatory versus home blood pressure monitoring. J Hum Hypertens. 2014 Apr;28(4):224-9. doi: 10.1038/jhh.2013.104. Epub 2013 Oct 24. PMID 24152822